CLINICAL TRIAL: NCT00016887
Title: Treatment of Mantle Cell Lymphomas at Advanced Stages: Prospective Randomized Comparison of Myeloablative Radiochemotherapy Followed by Blood Stem Cell Transplantation Versus Maintenance With Interferon Alpha in First Remission After Initial Cytoreductive Chemotherapy With an Anthracycline Containing Combination
Brief Title: Chemotherapy Followed by Radiation Therapy and Peripheral Stem Cell Transplant Compared With Chemotherapy Plus Interferon Alfa in Treating Patients With Stage III or Stage IV Mantle Cell Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: German Low Grade Lymphoma Study Group (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); Gruppo Italiano Studio Linfomi (Other); Lymphoma Study Association (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068609; GER-LGLSG-INTERGROUP-20995; EORTC-20995; GELA-INTERGROUP-20995; GISL-INTERGROUP-20995
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2003-08

CONDITIONS: Lymphoma
Keywords: stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Filgrastim; Interferon-alpha; Carmustine; Cyclophosphamide; Cytarabine; Dexamethasone; Etoposide; Melphalan; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interferon alfa
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: etoposide
Drug: melphalan
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill cancer cells. Peripheral stem cell transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Interferon alfa may interfere with the growth of cancer cells. It is not yet known whether giving more than one drug (combination chemotherapy) with radiation therapy and peripheral stem cell transplant is more effective than chemotherapy followed by interferon alfa in treating mantle cell lymphoma.

PURPOSE: This randomized phase III trial compares how well chemotherapy followed by radiation therapy, chemotherapy, and peripheral stem cell transplant works compared to chemotherapy plus interferon alfa in treating patients who have stage III or stage IV mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free survival of patients with previously untreated advanced mantle cell lymphoma treated with intensified chemotherapy followed by myeloablative radiochemotherapy and peripheral blood stem cell transplantation (PBSCT) vs standard therapy and interferon alfa maintenance.
* Compare the overall survival of patients treated with early vs late myeloablative radiochemotherapy and PBSCT.
* Compare disease-free survival and overall survival of patients treated with this regimen vs historic controls of similar cases.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to risk factors (ECOG performance status greater than 1, LDH serum level above normal, and/or extranodal lymphoma involvement) and participating center. Patients are randomized to 1 of 2 treatment arms.

* Induction: All patients receive 4 courses of cytoreductive chemotherapy comprising an anthracycline-containing combination. Patients not achieving complete remission after 4 courses receive 2 additional courses of induction chemotherapy. Patients without at least a partial response after 6 courses discontinue treatment; those with at least a partial response proceed to arm I or II.

Arm I

* Consolidation: Patients achieving complete or partial remission after 4-6 courses of induction therapy begin intensified chemotherapy within 6 weeks. Patients receive oral dexamethasone daily on days 1-10, carmustine IV on day 2, melphalan IV on day 3, etoposide IV daily and cytarabine IV twice a day on days 4-7. Patients also receive filgrastim (G-CSF) beginning on day 11 and continuing until peripheral blood stem cells (PBSC) are harvested.
* Within 4-6 weeks after PBSC harvest, patients undergo myeloablative radiochemotherapy comprising radiotherapy on days -6 to -4 and cyclophosphamide IV on days -3 to -2. Patients then undergo PBSC transplantation on day 0.

Arm II

* Consolidation: Patients receive 2 additional courses of induction chemotherapy as consolidation (for a total of 8 chemotherapy courses).
* Maintenance: Within 4 weeks after arm II consolidation, patients receive interferon alfa subcutaneously (SC) 3 days a week in the absence of unacceptable toxicity or disease progression or relapse. Patients who experience first relapse or progression during maintenance therapy may receive intensified chemotherapy as in arm I.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 210 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III or IV mantle cell lymphoma

  * Previously untreated
* Not qualified for primary potentially curative radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 to 65 years

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No impairment of liver function (unless due to lymphoma)
* Transaminases no greater than 3 times normal
* Bilirubin no greater than 2.0 mg/dL

Renal:

* No renal insufficiency
* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No manifest heart failure or coronary heart disease
* No severe uncontrolled hypertension

Pulmonary:

* No chronic lung disease with hypoxemia

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No severe uncontrolled diabetes mellitus

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior interferon
* No prior organ, bone marrow, or peripheral blood stem cell transplantation

Chemotherapy:

* No prior cytostatic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hiddemann, MD, PhD, Study Chair — Klinikum der Universitaet Muenchen - Grosshadern Campus; J. C. Kluin-Nelemans, MD, PhD, Study Chair — University Medical Center Groningen; Alessandro Levis, MD, Study Chair — Ospedale Civile Alessandria; Achiel Van Hoof, MD, Study Chair — AZ Sint-Jan
Locations (2):
- AZ Sint-Jan, Bruges, Belgium
- Ospedale Civile Alessandria, Alessandria, Italy

REFERENCES:
- [Derived] Determann O, Hoster E, Ott G, Wolfram Bernd H, Loddenkemper C, Leo Hansmann M, Barth TE, Unterhalt M, Hiddemann W, Dreyling M, Klapper W; European Mantle Cell Lymphoma Network and the German Low Grade Lymphoma Study Group. Ki-67 predicts outcome in advanced-stage mantle cell lymphoma patients treated with anti-CD20 immunochemotherapy: results from randomized trials of the European MCL Network and the German Low Grade Lymphoma Study Group. Blood. 2008 Feb 15;111(4):2385-7. doi: 10.1182/blood-2007-10-117010. Epub 2007 Dec 12. PMID 18077791